CLINICAL TRIAL: NCT06425679
Title: Cost-effectiveness and Efficacy of Physical Exercise on Mental and Physical Health in Older Adults: Role of Motivational Strategies and Digital Technology
Brief Title: Cost-effectiveness and Efficacy of Different Physical Exercise Interventions (ExerMOT4Health)
Acronym: ExerMOT4Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Instituto de investigación e innovación biomédica de Cádiz (Other); Universidad de Almeria (Other); Ministerio de Ciencia e Innovación, Spain (Other Government); State Research Agency, Spain (Other Government); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Ana Carbonell Baeza, PhD, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PID2021-123688OB-C31
Record Dates: First submitted 2024-04-26; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Physical Inactivity; Healthy Aging; Older Adult
Keywords: Aging; Exercise; Physical activity; Supervised; Home-based; Multidomain training; Multicomponent training; Physical health; Mental health; Quality of life; Physical function; Cost-effectiveness
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Supervised synchronous online exercise intervention without motivational strategies (Experimental)
  Interventions: Behavioral: Supervised synchronous online exercise intervention without motivational strategies
- Supervised synchronous online exercise intervention with motivational strategies (Experimental)
  Interventions: Behavioral: Supervised synchronous online exercise intervention with motivational strategies
- Supervised face to face exercise intervention without motivational strategies (Experimental)
  Interventions: Behavioral: Supervised face to face exercise intervention without motivational strategies
- Supervised face to face exercise intervention with motivational strategies (Experimental)
  Interventions: Behavioral: Supervised face to face exercise intervention with motivational strategies
- Control group (No Intervention): Participants will be advised to maintain their usual lifestyle.

INTERVENTIONS:
Behavioral: Supervised synchronous online exercise intervention without motivational strategies — Participants will carry out an online synchronic supervised physical exercise intervention through their computer/tablet or mobile phone at home. The exercise professional will supervise the participant's execution online. The training program comprises the same exercise structure and is based on the same muscle groups and movements as the supervised face to face groups. The exercise program will be divided into 3 different levels, progressing the difficulty every 8 weeks.. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises, 2 aerobic exercises, and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks
  Arms: Supervised synchronous online exercise intervention without motivational strategies
Behavioral: Supervised synchronous online exercise intervention with motivational strategies — Participants will carry out an online synchronic supervised physical exercise intervention through their computer/tablet or mobile phone at home. The exercise professional will supervise the participant's execution online and will also apply motivational strategies based on self-determination theory. The training program comprises the same exercise structure and is based on the same muscle groups and movements as the supervised face to face groups. The exercise program will be divided into 3 different levels, progressing the difficulty every 8 weeks. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises, 2 aerobic exercises, and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks.
  Arms: Supervised synchronous online exercise intervention with motivational strategies
Behavioral: Supervised face to face exercise intervention without motivational strategies — Participants will attend the sports facilities and perform the training in small groups, being supervised by an exercise professional. The training program comprises the same exercise structure and is based on the same muscle groups and movements as the online synchronic supervised groups, but is performed in a sports center. The exercise program will be divided into 3 different levels, progressing the difficulty every 8 weeks. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises, 2 aerobic exercises and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks.
  Arms: Supervised face to face exercise intervention without motivational strategies
Behavioral: Supervised face to face exercise intervention with motivational strategies — Participants will attend the sports facilities and perform the training in small groups, being supervised by an exercise professional who will also apply motivational strategies. The training program comprises the same exercise structure and is based on the same muscle groups and movements as the online synchronic supervised groups, but is performed in a sports center.
  The exercise program will be divided into 3 different levels, progressing the difficulty every 8 weeks. Each level will contain 3 different sessions including 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises, 2 aerobic exercises and 6 flexibility exercises. This multicomponent training will be performed 3 times per week (60 min/session) for 24 weeks.
  Arms: Supervised face to face exercise intervention with motivational strategies

SUMMARY:
Online exercise has increased in popularity during the pandemic, but there is no evidence of its feasibility and benefits in older people and the influence of motivational strategies. The main aims of this project are: i) To analyze the influence of applying or not motivational strategies during different physical exercise interventions (face-to-face and online) on the effect on mental health, physical health and adherence, according to sex/gender; ii) To analyze and compare the cost-effectiveness and efficacy of face-to-face and online exercise interventions on mental health, physical health and adherence, according to sex/gender. Participants will be 104 community-dwelling older adults (60-75 years) who will be randomized assigned to control, supervised face to face, supervised face to face plus motivation, synchronous online supervised exercise or synchronous online supervised exercise groups.

The control group will carry out the usual activities they have been doing, and the intervention groups will participate for 24 weeks in multicomponent exercise intervention. Study assessments will be made before starting the intervention, at the end and after 24 weeks of follow-up. Primary variables will be changes in mental and physical health, assessed by the Trail Making Test, the Yesavage Geriatric Depression Scale, and lower extremity power measured by the sit to stand test. Secondary outcomes will include other parameters of mental and physical health, blood markers, physical activity, and cost-effectiveness analysis. The dropout rate, the attendance at the sessions, the injuries and other adverse events suffered by the participants, and technical incidences produced in the online modality will also be recorded.

The results of this project will provide insight into the mental and physical health effects and feasibility of face-to-face and synchronous online supervised physical exercise interventions, and identify older adults' perceptions of the safety, barriers and facilitators of these interventions for future application and transfer to community settings.

DETAILED DESCRIPTION:
Scientific evidence has demonstrated the effects of multicomponent physical exercise on the mental and physical health of community-dwelling older people. Despite this, the interest of some older people in exercise is low and even a low percentage of older people practice it with sufficient frequency and intensity to obtain benefits in their mental and physical health. Recent studies have demonstrated the importance of using motivational strategies to generate adherence to exercise, but there are still no studies with community-dwelling older adults. Furthermore, the Covid-19 pandemic has shown that face-to-face physical exercise is not always possible, so it is necessary to have alternatives in case situations of social isolation and mobility restrictions return. It is also important to note that many older people have difficulty traveling to a sports center or living in rural environments, which makes it difficult to practice exercise regularly. Online exercise has increased in popularity during the pandemic, but there is no evidence of its feasibility and benefits in older people.

The specific aims of this study are:

1. To analyze the influence of applying or not motivational strategies during supervised face-to-face and synchronous online physical exercise interventions on the effect on mental health, physical health and adherence, according to sex/gender in the community setting.
2. To analyze and compare the cost-effectiveness and efficacy of supervised face-to-face and synchronous online exercise interventions vs usual lifestyle on mental health, physical health and adherence, according to sex/gender in the community setting, in short and long term (follow up).
3. To design and evaluate the feasibility of supervised face-to-face and synchronous online exercise interventions and to identify older adults' perceptions of safety, barriers and facilitators of supervised face-to-face and synchronous online physical exercise interventions for future application and transfer to the community setting.
4. To create audio-visual resources that explain how to implement safe face-to-face and synchronous online supervised physical exercise interventions in older men and women that promote adherence, based on scientific evidence, in the community setting.

Participants (N=104 community-dwelling older adults aged 60-75 years) will be randomized assigned to: 1) control, 2)supervised face to face, 3) supervised face to face plus motivation, 4) synchronous online supervised exercise or 5) synchronous online supervised exercise groups.

The control group will carry out the usual activities they have been doing, and the intervention groups will participate for 24 weeks in 3 sessions/week of multicomponent exercise intervention, being performed from home (online groups) or at a sport center, according to the assigned group. Each session will last 60 minutes and will include 10 warm-up and joint mobility exercises, 1 balance exercise, 7 strength exercises, 2 aerobic exercises, and 6 flexibility exercises.

Study assessments will be made before starting the intervention, at the end and after 24 weeks of follow-up. Primary variables will be changes in mental and physical health, assessed by the Trail Making Test, the Yesavage Geriatric Depression Scale, and lower extremity power measured by the sit-to-stand test. Secondary outcomes will include other parameters of mental and physical health, blood markers, physical activity, and cost-effectiveness analysis. We will also record the dropout rate, the attendance at the sessions, the injuries and other adverse events suffered by the participants, and technical incidences produced in the online modality.

ELIGIBILITY:
Inclusion Criteria:

* People from both sexes aged 60-75 years.
* Not to have diseases and disabilities that limit to be part of exercise interventions or avoid measurements.
* Not perform supervised moderate to vigorous physical activity >30 minutes and >3 days/week.
* To be able to communicate without problems.
* To be able to read and understand the aim of the project and informed consent form.
* To have a smartphone, tablet or computer with internet connection.

Exclusion Criteria:

* Acute or terminal illness.
* Myocardial infarction, coronary artery bypass grafting, angioplasty, angina, or other cardiac conditions in the past year.
* Uncontrolled medical problems that the general practitioner considers would preclude patients from undertaking the exercise program (e.g., acute systemic illness such as pneumonia, acute rheumatoid arthritis, and acute or unstable heart failure).
* Conditions requiring a specialized physical exercise program (e.g., uncontrolled epilepsy, significant neurological disease or impairment, inability to maintain an upright seated position or unable to move independently, multiple sclerosis, cancer, Parkinson's, Alzheimer's, or chronic obstructive pulmonary disease).
* General practitioner-diagnosed hypertension that has not been controlled.
* Uncontrolled Type I or Type II Diabetes.
* History of major psychiatric illness including schizophrenia, generalized anxiety disorder, or depression according to the DSM-5.
* Three or more self-reported falls in the last year.
* Not wanting to complete the study or be assigned to the control group;
* Be participating in another research study that may influence this project.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Performance | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  The Trail-Making Test Part A and B will be administered. Part A is based on number sequencing, participants link numbers from 1 to 25 in ascending order. Part B focuses on alternating numbers and letters in ascending order. The completion time will be registered in seconds (the lower duration, the best performance).
Depression | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  The short 15-item version of the Yesavage Geriatric Depression Scale will be used. This is a questionnaire used to screen for depression in older people. This scale consists of 15 items with a yes/no answer pattern, being the minimum score 0 and the maximum 15. The cut-off point for Depression is 5 or more.
Lower-body muscular function | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  Lower limb muscle performance will be assessed using the 30-seconds Chair Sit to Stand (30-s CST) test. The number of standing up in 30 seconds will be counted. A higher score, better performance.

SECONDARY OUTCOMES:
Upper-body muscular function | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  Grip strength will be measured with a digital hand-held dynamometer on both arms (Takei TKK5401, Tokyo, Japan).
  The test was performed in both standing and sitting positions, in both cases with the arm fully extended. A higher score, better performance.
Maximum walking speed (3, 4, 6 and 10-m) | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Maximum gait speed will be evaluated by measuring the time used to walk 3, 4, 6 and 10 meters linear distance at maximum pace without running. Gait speed is calculated by dividing the distance into registered walking time. A higher speed (or lower registered time) better performance.
Usual walking speed (3, 6 and 10-m) | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Usual gait speed will be evaluated by measuring the time used to walk 3, 6 and 10 meters linear distance at usual pace. Gait speed is calculated by dividing the distance into registered walking time. A higher speed (or lower registered time) better performance.
Short Physical Performance Battery (SPPB) | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  It consists of three parts: the ability to stand with feet together in side-to-side, semi-tandem, and tandem positions (balance), 4-meters walk test (speed), and 5 times sit-to-stand (muscle power). Each part is scored from 0 to 4, with a total SPPB score of 12 points, a higher score, better performance.
Senior Fitness Test (SFT) | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  SFT battery includes 30-second chair stand test (lower-body strength), 30-second arm curl test (upper-body strength), 6-minute walk test (aerobic endurance), Chair sit-and-reach test (lower-body flexibility), Back scratch test (upper-body flexibility) and 8-foot up-and-go test (agility and dynamic balance).
Resting blood pressure | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  Systolic and diastolic blood pressure will be assessed in a seated position, twice, 2 minutes apart, after 5 minutes at rest, using a digital upper arm blood pressure monitor (OMRON M6, Spain). Blood pressure will be assessed at the level of the right atrium, with the participant's back supported and uncrossed legs with both feet on the floor.
Resting heart rate | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  Heart rate will be assessed in a seated position twice, 2 minutes apart, after 5 minutes at rest, units will be bpm (beats per minute), using a digital upper arm blood pressure monitor (OMRON M6, Spain).
Anthropometry | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Height will be measured with a stadiometer (Seca 213, Hamburg, Germany). Body mass will be measured using a body composition analyzer (InBody 770, Biospace, California, USA). The participant will be barefoot and wearing as minimally clothed as possible.
  Body mass index will be calculated as body mass (kg) divided by height (m) squared (kg·m-2).
Body perimeters | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Waist and hip perimeters will be measured in upright position in accordance with the ISAK guidelines with a circumference tape (Lukfin, W606PM) following the standardized protocol, as well as calf perimeter in a sitting position.
Body composition | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  Body Composition will be measured using a body composition analyzer (InBody 770, Biospace, California, USA), following the standardized protocol. Fat mass (kg and %), fat free mass (kg and %) and skeletal muscle mass (kg and %) will be obtained.
Health-related quality of life | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  The EuroQol-5D questionnaire will be used for assessing the health-related quality of live of the participants, including five dimensions and a visual analogue scale. The 5 dimensions included in the descriptive system are (1) mobility, (2) self-care, (3) usual activities, (4) pain/discomfort, and (5) anxiety/depression. Responses will be coded according to the three-level scale for each dimension. A utility value will be assigned to each combination of responses. This index provides a quantitative measure of each individual's health-related quality of life, where 0 represents the worst possible health and 1 represents the best possible health.The EQ-VAS scale consists of asking participants to indicate their current health status from 0 ("worst imaginable health status") to 100 ("best imaginable health status").
Cognitive Performance- The Montreal Cognitive Assessment | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The Montreal Cognitive Assessment (MoCA) assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score ranged from 0 to 30, and the highest score indicates better performance.
Cognitive Performance-The Stroop Color and Word Test (SCWT) | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The Stroop Color and Word Test (SCWT) is divided into three conditions, the first condition consists of reading color names printed in black ink, in the second condition the participant will read colors printed in an "X", and the third condition consists of naming the ink color instead of reading the word. All conditions contain 100 words, and time is limited to 45 seconds for each condition. The total number of correct words for each condition will be recorded, indicating that the higher the number of correct words, the better the performance.
Cognitive Performance- Digit Span test of the Wechsler Adult Intelligence Scale III | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Digit Span test of the Wechsler Adult Intelligence Scale III (WAIS III). Participants will be asked to recall a list of numbers in the order given (forward or backwards). The test is finished when for the same item, the participant fails two attempts. A total number of correct answers will be registered for each condition, ranging from 0 to 30, with the highest scores being the best performance.
Cognitive Performance-Clock Drawing Test (CDT). | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The test consists of drawing a clock with a given time (11:10). The total score is the sum of the scores given to dial, numbers and clock faces, ranging from 0 to 10 with the highest scores being the best performance.
Cognitive Performance- Digit Symbol Substitution Test | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Digit Symbol Substitution Test. The participant will fill in a series of coded symbols for 90 and 120 seconds. The total number of responses as well as errors are recorded. In this test, the higher the score, the better the performance.
Anxiety | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  The Zung Anxiety Self-Assessment Scale will be used to assess anxiety symptoms. It consists of 20 items with a 4-point response scale ranging from 1 (not at all or hardly ever) to 4 (most or all of the time), obtaining a maximum score of 80. The higher the score, the higher anxiety.
Physical activity and sedentary behavior patterns assessed by accelerometry. | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Physical activity and sedentary behavior will be assessed by accelerometry ((Actigraph GT3X, MTI, USA). The devices will be placed on the subject's non-dominant wrist using a watch strap for 8 days.
Physical activity and sedentary behavior patterns by questionnaire | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Physical activity and sedentary behavior will be assessed by the International Physical Activity Questionnaire-Short form (IPAQ). This questionnaire ask about the time spent on vigorous, moderate, walking and sitting activities in the last 7 days.
Sleep assessed by accelerometry | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The number of hours of sleep will be assessed by accelerometry ((Actigraph GT3X, MTI, USA). The devices will be placed on the subject's non-dominant wrist using a watch strap for 8 days.
Sleep assessed by questionnaire | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  The Pittsburgh Sleep Quality Index consists of 19 self-assessed questions and 5 partner-assessed questions. The 19 items are combined to form seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction), each with a range of 0 to 3 points. The total score ranges from 0 to 21, where 0 points represents no difficulties and 21 points represents severe difficulties and worse sleep quality.
Serum BDNF | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Blood samples will be collected in the morning after an overnight fast and at least 24 h after the last exercise session. After collection, tubes will be centrifuged at 3500 rpm for 10 min. Serum obtained for each participant will be stored in aliquots at -80 °C until analysis. Serum BDNF (ng/mL) will be quantified using a sandwich enzyme-linked immunosorbent assay (ELISA). Human BDNF Quantikine Immunoassay (R&D Systems, Minneapolis, MN) will be performed according to the manufacturer's instructions.
Serum α-Klotho | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Blood samples will be collected in the morning after an overnight fast and at least 24 h after the last exercise session. After collection, tubes will be centrifuged at 3500 rpm for 10 min. Serum obtained for each participant will be stored in aliquots at -80 °C until analysis. A commercial enzyme-linked immunosorbent assay (ELISA) will be performed to measure α-klotho serum concentration (pg/ml) according to the manufacturer's protocol (Human soluble α-Klotho Assay Kit JP27998, Immuno-Biological Laboratories Co., Ltd., Gunma, Japan). The quantification will be performed spectrophotometrically using a FLUOstar OPTIMA Microplate Reader (ThermoFisher Scientific, Waltham, MA, USA) and Optima Control software version 2.20.
Routinary blood serum analysis | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Glucose, uric acid, urea, creatinine, bilirubin, sodium, potassium, chloride, calcium, phosphorus, total proteins, albumin, cholesterol, cholesterol-HDL, cholesterol-LDL (calculated), triglycerides, aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyltransferase (GGT),alkaline phosphatase, lactate dehydrogenase (LDH), creatine kinase (CK,) will be measured using routinary clinical techniques.
Hemogram | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  It consists of the analysis following parameters: red blood cell count, hemoglobin concentration, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red cell distribution width, white blood cell count, differential white blood cell count, platelet count and mean platelet volume
Motivators and barriers to exercise | Baseline (week 0), post-intervention (week 25), and follow-up (week 48).
  Motivators and barriers to exercise will be measured using the Exercise Benefits/Barriers Scale. It is a 43-item instrument with a four-response Likert-type scale; Twenty-nine items are related to the benefits, while the remaining 14 are barriers. - The total score of the instrument can range from 43 to 172 points, with higher scores indicating a more positive perception of exercise.
Motivation to exercise according to self-determination theory | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  The Behavioral Regulation during Exercise Questionnaire (BREQ-3) comprises 23 items (4 for intrinsic regulation, 4 for integrated regulation, 3 for identified regulation, 4 for introjected regulation, 4 for external regulation and 4 for amotivation) that measure the stages of the self-determination theory with respect to motivation to exercise. Participants will answer each item on a 5-point scale ranging from 0 (not true for me) to 4 (very true for me). Higher scores on identified regulation, integrated regulation and intrinsic motivation are generally considered indicative of a more self-determined and healthy motivation towards exercise. On the other hand, higher scores on amotivation, external regulation and introjected regulation generally indicate less self-determined motivation.
Basic Psychological Needs in Exercise | Baseline (week 0), Post-intervention (week 25) and follow-up (week 48)
  The Basic Psychological Needs in Exercise Scale (BPNES) is composed of 12 items assessing the satisfaction of the three basic psychological needs in physical exercise contexts: competence, autonomy and relationship with others. A 5-point likert scale is used: (1) Do not agree at all, (2) Somewhat agree, (3) Somewhat agree, (4) Strongly agree, and (5) Strongly agree.using : (1) I don't agree at all, (2) I agree a little bit, (3) I somewhat agree, (4) I agree a lot, and (5) I completely agree. For each need, a minimum score of 4 points and a maximum of 20 points can be obtained. The score for the total questionnaire would be a minimum of 12 points and a maximum of 60 points. A higher score reflects a better satisfaction of basic psychological needs.
Satisfaction with Life | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  The Satisfaction with Life Scale is a 5-item instrument with a Likert-type scale ranging from 1 to 5 points, and measures overall subjective happiness through statements in which participants rate themselves. The higher the score, the higher the satisfaction with life.
Sociodemographic characteristics questionnaire | Baseline (week 0), post-intervention (week 25), and follow-up (week 48)
  Age, sex, marital status, educational level, socioeconomic status, employment status, self-rated health, family history of Alzheimer, pathologies diagnosed, number of falls during the previous year, consumption of medicines, and tobacco and alcohol consumption will be determined by this questionnaire
Cost-Effectiveness Analysis | Through intervention completion (24 weeks)
  A cost-effectiveness analysis will be performed to assess the expenses associated with each intervention group, utilizing the EQ-5D questionnaire to evaluate changes in health states.The analysis will focus on the following key metrics, the Quality-Adjusted Life-Year (QALY) and the Incremental Cost-Effectiveness Ratio (ICER).
  The Cost-Utility analysis examines an intervention's cost-effectiveness by considering expenses and the impact on patients' quality of life. QALYs provide a comprehensive measure of both the quantity and quality of life, calculated by multiplying the utility weights assigned to each health state by the time spent in that state. The cost per QALY gained is determined by dividing the total intervention costs by the total QALYs gained.
  The ICER compares the cost-effectiveness of two interventions by evaluating the difference in costs and effects (QALYs gained). A positive ICER indicates that Intervention A is more expensive and less effective than Intervention B
Adherence to physical training program | Through intervention completion (week 24)
  Adherence to physical training program will be recorded by the trainers. It will be calculated as a percentage ([sessions completed/total sessions expected] x 100), where 0 % indicates total non-adherence and 100 % indicates full adherence to the exercise intervention.
Exercise during follow-up period | Follow-up (week 48)
  During the 24-week follow-up, the investigators will assess through an ad-hoc self-reported questionnaire whether or not participants exercised during the follow up period (24 weeks), the exercise modality performed, if the exercise was supervised center-based and/or unsupervised/supervised home-based, the number of weekly exercise sessions performed, the average time and the subjective intensity perceived (light, moderate or vigorous).
Falls and adverse events | Through intervention completion (24 weeks)
  Participants in the supervised synchronous online exercise and control groups will record in a diary their falls and adverse events during and outside exercise sessions. In the supervised face to face groups, supervisors will register the incidence of falls during exercise sessions an participants will register them outside the exercise sessions using the diary.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carbonell Baeza, PhD, Principal Investigator — University of Cadiz; Pablo Jorge Marcos Pardo, PhD, Principal Investigator — Universidad de Almeria
Locations (2):
- Spain (2):
  - Universidad de Almeria, Almería, Almeria
  - University of Cadiz, Puerto Real, Cadiz

IPD SHARING:
Plan to Share IPD: No